CLINICAL TRIAL: NCT06646666
Title: Efficacy and Safety of All-trans Retinoic Acid (ATRA)-Based Chemo-free Bridging/Maintenance Therapy in CAR-T Treatment of High-risk Relapsed/Refractory B-NHL Ineligible for High-dose Chemotherapy （HDCT） and Autologous Stem Cell Transplantation （ASCT）
Brief Title: ARTA-based Chemo-free Bridging/Maintenance Therapy in CAR-T Treatment for High-Risk R/R B-NHL Ineligible for HDCT and ASCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T 002
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Tretinoin; zanubrutinib; Radiotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARTA-based Chemo-free bridging therapy to CAR-T and maintenance therapy post CAR-T (Experimental)
  Interventions: Drug: All-trans retinoic acid; Drug: zanubrutinib; Radiation: radiotherapy; Drug: CAR-T; Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: All-trans retinoic acid — 10mg，tid，po (After apheresis and continued until post-infusion)
Drug: zanubrutinib — 160mg，bid，po (prior to apheresis and continued until post-infusion)
Radiation: radiotherapy — If the patient's specific lesions are suitable for radiotherapy
Drug: CAR-T — CAR-T cell therapy
Drug: PD-1 inhibitor — IV 200 mg on D1, Q3W

SUMMARY:
This is a single-center, open-label, prospective study enrolling high-risk (tumor diameter > 4 cm) relapsed/refractory B-NHL patients ineligible for HDCT and ASCT. The treatment consists of ATRA combined with zanubrutinib ± radiotherapy and CAR-T therapy. Based on the efficacy at day 28 post-CAR-T infusion, patients achieving CR will receive 3 months of ATRA and zanubrutinib, while those with PR will receive 3 months of zanubrutinib plus 2 years of ATRA and a PD-1 inhibitor. Patients with stable disease or progression will discontinue. The primary endpoint is the 3-month CR rate following CAR-T infusion.

ELIGIBILITY:
Inclusion Criteria:

* Willingly sign the informed consent form.
* Age ≥ 18 years, any gender.
* Histologically confirmed as B-cell non-Hodgkin lymphoma, including:

  * Diffuse large B-cell lymphoma (DLBCL) not otherwise specified (DLBCL-NOS)
  * Transformed follicular lymphoma (tFL)
  * High-grade B-cell lymphoma (HGBL) with MYC, BCL2, and/or BCL6 rearrangements
  * High-grade B-cell lymphoma not otherwise specified (HGBL-NOS)
  * Primary mediastinal large B-cell lymphoma (PMBL)
  * Follicular lymphoma grade 3b (FL3b)
* Patients must have experienced at least one line of treatment for relapsed or refractory disease, meeting the following definitions:

  * Refractory: At least partial response (PR) after the last chemotherapy or relapse within 12 months after autologous transplantation.
  * Relapsed: Complete response (CR) after the last chemotherapy, followed by relapse before enrollment, or relapse or progression 12 months or longer after autologous transplantation.
* Maximum tumor diameter (long axis) > 4 cm.
* Evaluator determines that the patient does not meet HDCT/ASCT criteria and meets at least one of the following:

  * Age ≥ 60 years
  * ECOG score = 2
  * FEV1% or DLCO% ≤ 60%
  * LVEF < 50%
  * Creatinine clearance < 60 mL/min
  * ALT or AST > 2× upper limit of normal (ULN)
  * Patient unwilling to receive high-dose chemotherapy and autologous stem cell transplantation.
* Measurable target lesions: lymph nodes ≥ 15 mm in longest diameter, or extranodal lesions > 10 mm.
* Expected survival ≥ 12 weeks.
* Laboratory tests must meet the following requirements at screening:

  * Lymphocyte count ≥ 0.1 × 10^9/L
  * Hemoglobin ≥ 80 g/L
  * Platelets ≥ 50 × 10^9/L
  * ALT/AST ≤ 5 × ULN and total bilirubin < 2 × ULN
  * Creatinine clearance ≥ 30 mL/min
  * Lung function: ≤ CTCAE grade 1 dyspnea, and oxygen saturation (SpO2) ≥ 92% in room air.
  * LVEF ≥ 40%
* Patients with primary central nervous system lymphoma are allowed (secondary CNS lymphoma is not allowed).
* Sufficient venous access for apheresis, and no other contraindications for blood cell separation; female participants of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* History of allergy to any component of the cellular product or study treatment.
* History of allogeneic hematopoietic stem cell transplantation.
* History of organ transplantation.
* Patients with active viral hepatitis requiring treatment, including:

  * Chronic HBV carriers with HBV DNA ≥ 500 IU/mL.
  * Positive HCV RNA in patients with positive HCV antibodies.
  * Positive HIV antibodies (HIV-Ab).
  * Positive Treponema pallidum antibodies (TP-Ab).
  * Elevated CMV DNA or EBV DNA above normal limits.
* Clinical significance of CNS diseases
* Presence of active primary central nervous system lymphoma.
* Prior treatment with other genetically modified T-cell therapies or CAR-T therapies.
* Severe genetic diseases or autoimmune diseases (e.g., systemic lupus erythematosus).
* Thromboembolic events (e.g., myocardial infarction, pulmonary embolism, deep vein thrombosis) within 6 months prior to screening.
* History of malignancies other than the indication for this trial within the last 5 years, except for in situ cancers (e.g., cervical, bladder, breast) or non-melanoma skin cancer.
* Active infections requiring systemic treatment or uncontrolled infections.
* Received lenalidomide, calcineurin inhibitors, chemotherapy (e.g., methotrexate, cyclophosphamide, ifosfamide, nitrogen mustard, or melphalan), mycophenolate, thalidomide, immunosuppressive antibodies (e.g., anti-TNF, anti-IL6, or anti-IL6R), radiation therapy, or any drug that binds FKBP12 (e.g., rapamycin, tacrolimus, everolimus) within 4 weeks prior to PBMC collection.
* Pregnant or breastfeeding women, or men or women of childbearing potential unwilling to use contraception during the trial and for 2 years after RJ CAR-T 002 cell infusion.
* Participation in other drug clinical trials (e.g., new drug trials, registrational studies, investigator-initiated trials) within 4 weeks prior to PBMC collection.
* Researcher's judgment that the patient is unsuitable for the trial (e.g., poor compliance, drug abuse).
* Vaccination with live or attenuated vaccines within 3 months prior to PBMC collection, or expected vaccination during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate at 3-month | 3 months post CAR-T infusion
  Complete response rate at 3-month is defined as the incidence of subjects achieving complete remission (CR) within 3 months after CAR-T infusion according to the Lugano Classification (Cheson et al, 2014), as determined by study investigators.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years post CAR-T infusion
  PFS is defined as the time from the CAR-T infusion date to the date of disease progression or death from any cause.
Overall Survival (OS) | 2 years post CAR-T infusion
  OS is defined as the time from CAR-T infusion to the date of death from any cause.
Adverse Events rate as assessed by CTCAE version 5.0 | 2 years post CAR-T infusion
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Shanghai Institute of Hematology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China